CLINICAL TRIAL: NCT06275282
Title: Regenerative Peripheral Nerve Interfaces to Enhance Function and Sensation in People With Transfemoral Amputation
Brief Title: Regenerative Peripheral Nerve Interface for Control of Lower Limb Prostheses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Deanna H Gates, Professor, School of Kinesiology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00235849
Record Dates: First submitted 2024-02-09; First posted 2024-02-23 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Amputation; Prostheses and Implants
Keywords: RPNI; Regenerative Peripheral Nerve Interface; Implanted Electrodes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Regenerative Peripheral Nerve Interface (RPNI) (Experimental): Participants will have regenerative peripheral nerve interfaces (RPNIs) created on nerves in their residual thighs. During either the same surgery or a separate surgery, electrodes will be implanted into these RPNIs.
  Interventions: Device: Intramuscular electrodes

INTERVENTIONS:
Device: Intramuscular electrodes — Participants will have regenerative peripheral nerve interfaces (RPNIs) created on nerves in their residual thighs. During either the same surgery or a separate surgery, small electrodes will be implanted into these RPNIs.

SUMMARY:
Individuals with an above-knee lower limb amputation are known to walk more slowly, expend more energy, have a greater risk of falling, and have reduced quality of life compared to individuals without amputation and those with below knee amputation. One of the driving factors behind these deficits is the lack of active function provided by above-knee prostheses with prosthetic knees and ankles. While many prosthetic devices have been developed for functional restoration after major lower extremity amputation, there remains no stable interface to facilitate reliable, long-term volitional control of an advanced robotic limb capable moving multiple joints. Moreover, there is no existing interface that provides useful sensory feedback that in turn enhances the functional capabilities of the prosthesis. To achieve both greater signal specificity and long-term signal stability, we have developed a biologic interface known as the Regenerative Peripheral Nerve Interface (RPNI). An RPNI consists of a peripheral nerve that is implanted into a free muscle graft that would otherwise go unused in the residual limb. As the nerve grows, it reinnervates the free muscle graft which undergoes a predictable sequence of revascularization and regeneration.

The main questions it aims to answer are:

1. Can the amplitude, movement specificity and stability of sciatic nerve RPNI electromyography (EMG) signals be detected up to one year post RPNI surgery?
2. Do RPNIs contain information to enable control of a physical motorized prosthetic leg with multiple degrees of freedom?
3. Does stimulation of sciatic nerve RPNIs provides meaningful sensory feedback?

Consenting participants with unilateral transfemoral amputation (TFA) will:

1. Undergo RPNI surgery and electrode implantation in the residual limb.
2. Attend regular follow-up visits following surgery to assess the health and signal strength of the RPNIs and their ability to use a prescribed prosthesis between 3- and 12-months following implantation.
3. Undergo explantation of electrodes following the conclusion of data collection.

DETAILED DESCRIPTION:
Background: While many prosthetic devices have been developed for functional restoration after major lower extremity amputation, there is no stable interface to provide reliable, long-term volitional control of an advanced robotic limb capable of multiple degrees of freedom. Moreover, there is no existing interface that provides useful sensory feedback that in turn enhances the functional capabilities of the prosthesis. To address these limitations, the investigators propose use of a novel biologic interface known as the Regenerative Peripheral Nerve Interface (RPNI). An RPNI consists of a peripheral nerve that is implanted into a free muscle graft. As the nerve grows, it reinnervates the free muscle graft which undergoes a predictable sequence of revascularization and regeneration. The RPNI leverages these biological processes to provide three essential benefits to people with amputation: 1) intuitive motor control, 2) sensory feedback, and 3) reduction of post-amputation pain.

Objective/Hypotheses: The objective of this application is to (1) determine the extent to which the RPNIs enable generation of high-fidelity motor control signals for a powered knee-ankle prosthesis and (2) demonstrate that meaningful sensory feedback can be generated from stimulation of sciatic nerve RPNIs.

Specific Aims: The specific aims are to: (1) Evaluate the amplitude, movement specificity and stability of sciatic nerve RPNI electromyography (EMG) signals up to one year post RPNI surgery, (2) Assess functional movement performance using sciatic nerve RPNI signals for control of a physical motorized prosthetic leg with multiple degrees of freedom, and (3) Determine whether stimulation of sciatic nerve RPNIs provides meaningful sensory feedback.

Study design: This project is the first clinical investigation of RPNIs in people with lower-limb amputation. The study will recruit 3 individuals with transfemoral amputation. RPNIs will be surgically constructed on the sciatic nerve and intramuscular electrodes will be implanted into these RPNIs and residual muscles. Experiments will then be conducted at regular intervals up to one year post RPNI surgery. These experiments will measure the EMG signals generated by RPNIs in response to volitional movement of the phantom limb. These signals will then be used to control a two-joint powered prosthesis during cyclic and unpredictable movements. Functional movement, pain, and other patient-reported outcomes will be collected for data analysis. Additionally, RPNIs will be electrically stimulated to elicit sensation. Stimulation will also be provided during the performance of functional tasks.

At the completion of data collection, participants will undergo electrode explantation and complete a postoperative visit to assess recovery, pain and any associated adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral amputation of the leg proximal to the knee at least 6 months prior to enrollment.
* Low surgical risk (American Society of Anesthesiologists Class I and II).
* For participants without existing RPNI grafts (at the time of enrollment), the residual limb must have sufficient soft tissue quality to support performance of the RPNI operative procedures. Participants sustaining severe crushing or avulsion injuries with substantial superficial and deep scarring may not be appropriate candidates for inclusion in the study.
* Amputee Mobility Predictor with prosthesis (AMPPRO) score of at least 37 (Gailey et al. 2002).
* Sufficient clearance to a motorized prosthetic leg without the necessity for shoe lifts or extenders on the contralateral limb.

Exclusion Criteria:

* Severe pain syndrome including complex regional pain syndrome or severe phantom pain. All of these conditions would suggest pathological activity of the nerve and would exclude the participant from participation.
* Untreated mental health disorders and if they have any DSM-5 diagnoses, they must receive approval to participate from their mental health professional.
* Any medical conditions that, in the opinion of the Principal Investigator, would place them at high risk for a surgical procedure including recent myocardial infarction, cerebrovascular accidents, deep venous thrombosis, pulmonary embolus, uncontrolled diabetes, or end stage renal disease.
* Participants must not have used tobacco for at least one month prior to enrollment in the study.
* Participants must agree to not use tobacco for the duration of the study.
* Pregnancy.
* No other indwelling electronic implants like pacemakers, implantable cardioverter defibrillators, implantable neurostimulators, body worn insulin pumps, or body worn patient monitoring devices.
* Severe peripheral vascular occlusive disease, venous hypertension of the extremity, or severe lymphedema of the extremity.
* An autoimmune condition which is not well controlled by medication.
* A significant injury of the contralateral limb.
* Significant, uncorrected vision problems.
* Impaired mental capacity that negatively impacts verbal communication with the clinicians and research team or requires a Legally Authorized Representative to facilitate communication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain in residual and phantom limbs | through study completion, an average of 1 year
  Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity-Short Form 3a
Neuropathic Pain in residual limb | through study completion, an average of 1 year
  Leeds Assessment of Neuropathic Symptoms and Signs (LANSS)
Health-Related Quality of Life | through study completion, an average of 1 year
  Participants will complete the RAND 36-Item Short Form Health Survey (SF-36)
Amplitude and signal-to-noise ratio for each RPNI | Postoperatively at each experimental visit at 3,6,9 & 12 months
  Participants will be instructed to make large, sustained movements with their phantom lower extremity while in a seated position to estimate their maximum voluntary contraction. They will repeat this process five times for each movement. The signal-to-noise ratio (SNR) will be calculated as the ratio of that signal to the quiescent period signals.
Classification accuracy for movements of the phantom limb | Postoperatively at each experimental visit at 3,6,9 & 12 months
  Participants will move their phantom limb to match a virtual limb shown on a screen. We will measure how accurately we can predict the intended movement using muscle activity signals from RPNIs and residual muscles
Threshold for sensation after electrical stimulation of RPNI | Postoperatively at each experimental visit at 3,6,9 & 12 months
  We will stimulate RPNIs electrically through the implanted electrodes. We will quantify the charge necessary for the participant to feel sensation (perception threshold) and the minimum charge that becomes uncomfortable (discomfort threshold). We will also record the location and quality of the sensation felt at each threshold

CONTACTS AND LOCATIONS:
Overall Officials: Deanna Gates, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No